CLINICAL TRIAL: NCT02490865
Title: Systemic Bioactivity of Inhaled Nebulized RNS60
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08.1.2.H8
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Systemic Bioactivity of Nebulized RNS60
MeSH Terms: interventions — RNS60; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RNS60 (Experimental): Administration of nebulized RNS60 to test for systemic bioactivity
  Interventions: Drug: RNS60
- Normal Saline (Placebo Comparator): Administration of normal saline used as control
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: RNS60 — RNS60, 4 ml dose nebulized twice daily
  Arms: RNS60
Drug: Normal saline — Normal Saline, 4 ml dose nebulized twice daily
  Arms: Normal Saline

SUMMARY:
The study aims to determine the effects of nebulized RNS60 on selected biomarkers in the circulation.

DETAILED DESCRIPTION:
The study is a double-blind, placebo controlled, parallel design study. Participants will be randomized to receive 2 daily doses of either nebulised RNS60 or placebo (n=28 per group) for 22 days. On day 19 they will undergo an exercise protocol to induce muscle damage and blood samples will be taken on days 19, 20, 21 and 23 to determine the effects on CK and hsCRP. ROM and pain VAS assessments will also be completed.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
2. The participant has signed the ICF.
3. Healthy male or female participants aged 18-45 years inclusive. Attempts will be made to achieve an equal gender ratio through appropriate screening procedures, but a failure to do so will not preclude analysis of the final data set.
4. BMI between 19 and 27 kg/m2.
5. The participant is, in the opinion of the investigator, healthy on the basis of medical history and vital signs.
6. Available for follow-up for the duration of the study.
7. Non-smokers (no smoking or use of nicotine replacements (including e-cigarettes) in the previous month before screening or during the study)
8. Agree to abstain from donating blood during the study.
9. Men and women of reproductive potential who document use of adequate contraception during the study and for 1 month following the last day of treatment (Day 23)
10. Willing to refrain from taking anti-inflammatory medications during the study (particularly ibuprofen).

Exclusion Criteria:

1. Clinically significant psychiatric, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological (particularly myasthenia gravis), immunological, or haematological disease or abnormality, as determined by the study physician.
2. History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1.
3. History of significant musculoskeletal upper limb injury.
4. Participating in regular (≥ 2 times per week) upper body resistance exercise training within 6 weeks of Visit 1.
5. FEV1 < 80% or FEV1/FEC of < 75%
6. Use of steroids or immunosuppressive/immunomodulating drugs either orally or parenterally within 3 months of Visit 1.
7. Use of NSAIDs and other OTC medications within 2 weeks of Visit 1.
8. Use of any dietary/nutritional supplements, including vitamins and minerals, in the 2 weeks before Visit 1.
9. Positive urinary pregnancy test.
10. Pregnant or lactating at any point during the study from screening to final visit.
11. Following a weight reducing diet.
12. Currently participating in another clinical trial with an investigational or non-investigational drug or device, or has participated in another clinical trial within the 3 months preceding Visit 1.
13. Any condition that, in the investigator's opinion, compromises the participant's ability to meet protocol requirements or to complete the study.
14. Receipt of blood products or immunoglobin, within 3 months of visit 1.
15. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

No waivers from the Protocol will be allowed.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in serum concentration of creatine kinase (CK) | 4 days post exercise
Change in serum concentration of highly sensitive C-reactive protein (hsCRP) | 4 days post exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom